CLINICAL TRIAL: NCT00802971
Title: Prevalence of Idiopathic Reactive Hypoglycaemia and Impact of Fructo-Oligosaccharide Supplementation on Blood Glucose Variability
Brief Title: Idiopathic Reactive Hypoglycaemia and Treatment With Fructo-Oligosaccharide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Odd Erik Johansen, Odd Erik Johansen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRH - FOS
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Hypoglycemia
Keywords: Reactive hypoglycaemia; Fiber; Prevalence; Randomised controlled trial; Idiopathic reactive hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: FOS (Experimental): Oligofructose (FOS, BioCare Ltd, Birmingham, England) powder will be distributed in sachets of 10 g. Two sachets are to be included in daily nutrition, preferentially 10 g diluted in water at breakfast and before supper.
  Interventions: Dietary Supplement: FOS
- 2: Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: FOS — Oligofructose (FOS, BioCare Ltd, Birmingham, England) powder will be distributed in sachets of 10 g. Two sachets are to be included in daily nutrition, preferentially 10 g diluted in water at breakfast and before supper.
  Arms: 1: FOS

SUMMARY:
Idiopathic reactive hypoglycemia (IRH) describes a condition where recurrent episodes of symptomatic hypoglycemia occurs one to four hours after a meal, usually following meals rich in carbohydrates. Differential diagnoses to be excluded include those caused by isulinomas or bariatric surgery (dumping syndrome), or iatrogenic induced hypoglycaemia.

The prevalence of IRH is not fully known. A British trial among 1136 random chosen women aged 17-50, reported that 37.9% experienced symptomatic hypoglycemia four times every month (mean value). However, not all reported symptoms attributed to a low blood glucose (BG) correlates with measured low levels of BG and a "true" hypoglycaemic episode, i.e., as defined by American Diabetes Association (ADA) when plasma BG value is < 3,9 mmol/l with or without accompanying symptoms. This was underscored in three studies from England, Canada and Denmark, in whom all reported hypoglycaemic symptoms, but in whom accompanying plasma glucose values < 3,3 mmol/l during hypoglycaemic symptoms only occurred in 23, 47 and 0% of the study subjects, respectively. The majority of those with symptoms related to IRH hence are having these symptoms without being classified as hypoglycemic according to conventional interpretations. However, a new (2005) ADA definition; relative hypoglycemia, also comprise these symptomatic cases of hypoglycemia following a plasma glucose > 3,9 mmol/l.

Hormonal and cerebral mechanisms tightly control the complex interplay of mechanisms involved in regulating BG concentration. Explanations for IRH are centralized around increased insulin secretion/sensitivity and/or down regulated transcription of glucagon receptor or reduced glucagons sensitivity- and secretion. Others assess an overabundance of adrenaline and cortisol, witch is excreted at the nadir of the BS curve (venous plasma glucose between 3.6 and 3.9). The latter event, during which typical symptoms is characterized of anxiety, fatigue, irritability, palpitations, nervousness, tachycardia, tremor and sweat.

Today, treatment is limited to dietary recommendations of eating frequent meals of moderate size, reasonably high in protein, and with a low glycaemic load. These advices keep cerebral glucose concentration stable and prohibit neuroglycopenic symptoms like hunger, dizziness, tingling, blurred vision, difficulty in thinking, and faintness. Pharmacologic attempts in treating IRH involves diazoxide, metformin, α-glucosidase inhibitor, glitazones and somatostatin, however, none of these medications are specifically indicated for the condition.

Fiber is a class of carbohydrate resistant to hydrolytic digestion in the upper bowel but fermented in the colon by bacterially produced enzymes. It makes the rate of ventricular emptying increase and prolongs the bowel transit time; thus having a minimal impact on BG values. Inulin and oligofructose are composed of polymers of oligofructose having characteristic features different from other fibers because of their physiological and biochemical attributes. Found in a variety of edible fruit and vegetables, their fermentation produces short-chain fatty acids that acidify the colonic content. This stimulates selectively the growth of beneficial and potentially health-promoting bifidobacteria and reduces potential harmful colon bacteria. Acting as prebiotica, oligofructose induces changes in the colonic epithelium and in miscellaneous colonic functions, inter alia, enhances calcium and magnesium absorption, modulates endocrine as well as immune functions and affects the metabolism of lipids positively. The latter, being at a systemic level, may contribute to modulating lipogenesis and reducing triglyceridemia by partially impairing hepatic cholesterol synthesis.

FOS has not yet been investigated thoroughly as a possible stabilizer of blood glucose. However, several non-oligofructose studies, using a high-fiber diet, indicates reduced pre-prandial BG values, less hypoglycemic cases, glukosuri, total cholesterol, triglycerides, VLDL cholesterol and area under the curve (AUC) in a 24 hours measurement (every 2 hour) of BG and insulin concentration.

Clinical evaluation of safety of inulin and oligofruktose as dietary fiber has reported 20 g/day of oligofructose to be well tolerated. The various GI side effects identified include abdominal pain and bloating, flatulence and osmotic diarrhea.

Despite the fact that fiber intake is proven inversely related to hypoglycemic events, possible benefits of daily FOS-supplementation have not yet been investigated systematically in persons suffering of IRH. Given the estimated high prevalence of IRH it is in our aim to:

1. Study the prevalence and characteristics of subjects with IRH in a relevant Norwegian study population of 414 study participants.
2. Evaluating the effect of FOS supplementation on blood glucose variability.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Ideopathic reactive hypoglycaemia defined as 1h or 2h glucose valued during OGTT < 3.9 mmol/l or 1h or 2h glucose values during OGTT < fasting glucose

Exclusion Criteria:

* Diabetes mellitus, impaired glucose tolerance, other reason for reactive hypoglycaemia than ideopacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Oligofructose, ingested along with a meal, contributes to a postponed increase in blood glucose and stabilizes the glucose metabolism. | 4 weeks

SECONDARY OUTCOMES:
Impact of FOS on 24-hours interstitial glucose AUC | 4 weeks
With FOS after 2 weeks there will be proportionate less study participants qualified for IRH diagnosis after 3 and 4 hours OGTT | 4 weeks
FOS for 2 weeks alteres lipid values (total cholesterol, triglycerides, LDL cholesterol, and HDL cholesterol). | 4 weeks
Fos for 2 weeks alteres fasting serum insulin and fasting glucagon | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Odd Erik Johansen, MD, PhD, Study Chair — Asker and Baerum Hospital